PRINCIPAL INVESTIGATOR: Jing Wu, MD

**STUDY TITLE:** Phase I Trial of Zotiraciclib (TG02) Plus Dose-Dense or

Metronomic Temozolomide Followed by Randomized Phase II Trial of Zotiraciclib (TG02) plus Temozolomide versus Temozolomide alone in Adults with Recurrent

Anaplastic Astrocytoma and Glioblastoma

STUDY SITE: NIH Clinical Center

Cohort: Affected Patient

Consent Version: 06/01/2020

# WHO DO YOU CONTACT ABOUT THIS STUDY?

Principal Investigator: Jing Wu, M.D., PhD Tel: 240-760-6036 Email: jing.wu3@nih.gov

This consent form describes a research study and is designed to help you decide if you would like to be a part of the research study.

You are being asked to take part in a research study at the National Institutes of Health (NIH). Members of the study team will talk with you about the information described in this document. Some people have personal, religious, or ethical beliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). Take the time needed to ask any questions and discuss this study with NIH staff, and with your family, friends, and personal health care providers. Taking part in research at the NIH is your choice.

If the individual being asked to participate in this research study is not able to give consent to be in this study, you are being asked to give permission for this person as their decision-maker. The term "you" refers to you as the decision-maker and/or the individual being asked to participate in this research, throughout the remainder of this document.

# IT IS YOUR CHOICE TO TAKE PART IN THE STUDY

You may choose not to take part in this study for any reason. If you join this study, you may change your mind and stop participating in the study at any time and for any reason. In either case, you will not lose any benefits to which you are otherwise entitled. However, to be seen at the NIH, you must be taking part in a study or are being considered for a study. If you do choose to leave the study, please inform your study team to ensure a safe withdrawal from the research.

### WHY IS THIS STUDY BEING DONE?

This study will test an investigational drug called Zotiraciclib (TG02) citrate. An "investigational drug" is a drug that is being tested and is not approved for sale in the United States by the Food and Drug Administration (FDA). The purpose of this research study is to find out what effects (good and bad) Zotiraciclib (TG02) citrate has on you and your cancer. You will also receive temozolomide which is FDA approved and commonly used for recurrent high-grade astrocytoma.

This study has two parts: a phase I part and a phase II part. In the phase I part, the main purpose is to learn about the safety of the study drug, Zotiraciclib (TG02). The study

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2) Version Date: 06/01/2020




investigators have given Zotiraciclib (TG02) citrate to people in this study and found the highest dose of Zotiraciclib (TG02) citrate that people can tolerate when given in combination with temozolomide in two different treatment schedules. It was also found that one temozolomide treatment schedule was better than the other. However, we want to make sure that the highest dose that people tolerated is also the dose you need. Providing direct medical benefit to you is not the purpose of this part of the study.

In the phase II part, the dose of Zotiraciclib (TG02) in combination temozolomide chosen in phase 1 will be compared to temozolomide alone. The dosing schedule of temozolomide used in this part of the study will depend on the response to each phase I part. The purpose of this part of the study is to find out if Zotiraciclib (TG02) citrate in combination temozolomide is as effective as temozolomide alone for people with the brain tumors.

### WHY ARE YOU BEING ASKED TO TAKE PART IN THIS STUDY?

We are asking you to be in this study because you have a brain tumor that has progressed after your standard treatment.

### HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY?

Up to 152 participants will take part in this study. Up to 72 participants will be enrolled in the phase I part and up to 80 participants will be enrolled in the phase II part.

# **DESCRIPTION OF RESEARCH STUDY**

You will also be enrolled in the Neuro Oncology Branch Natural History protocol to assess molecular markers of your brain tumor. If you agree to be in this study, we will ask you to do the following things:

# **BEFORE YOU BEGIN THE STUDY**

Before you can start this protocol, we will do an evaluation to see if you are eligible to participate in this study. You may be enrolled in a screening study to determine your eligibility. This will include a physical examination and blood laboratory studies. You will also need to have an MRI of the brain if you have not had one in 14 days and an EKG will be done. We must also be certain we have complete information about your history any past treatments, including surgeries. You will need to provide surgical tissue samples from prior surgeries. Women who are capable of having children will have a pregnancy test. You cannot take part in this study if you are pregnant.

Any concerns you or your clinician may have can be further explored, and you may be referred to a specialist for further evaluation or treatment if necessary.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)




#### **DURING THE STUDY**

You will also complete a questionnaire about the severity of your symptoms and the interference these symptoms have in your daily life over the last 24 hours. You will complete this symptom burden questionnaire before you start study therapy and whenever you have a CT scan or MRI. You will also complete a questionnaire related to symptoms associated with treatment on day 2, 8, 14, 21, and 28 of each cycle as described in the study visit table below. These questionnaires related to symptoms associated with treatment will not be done for some patients.

#### PHASE I

If you are found to be eligible to take part in this study, you will receive Zotiraciclib (TG02) plus temozolomide by mouth. We need you to keep a diary of when you take the temozolomide and the Zotiraciclib (TG02) and any symptoms you may have. The nurse will give you a diary form for this purpose. Please bring it along with all of your study medication bottles with you to clinic when you come at the end of each cycle, even if they are empty.

As indicated above, two schedules of temozolomide in combination with Zotiraciclib (TG02) have been tested on this study. In order to clarify the dose of the favored schedule, we will test a small group of participants (up to 12). If you are in this group, you will receive the following doses:

Temozolomide dosing schedule

Temozolomide can be given in a schedule referred to as "dose dense". In this study, dose dense temozolomide is given as 125 mg/m2 for 7 days on and 7 days off in each cycle. In the phase I part of this study, participants will be assigned to receive Zotiraciclib (TG02) plus dose dense temozolomide (Arm 1).

Zotiraciclib (TG02) Dosing

You will take the first 200 mg dose of Zotiraciclib (TG02) 3 days prior to Day1 of cycle 1. You will take a 200 mg dose of Zotiraciclib (TG02) on days 1, 12, 15, and 26 of every 28-day cycle in all the cycles.

The 12 participants treated at the TG02 200 mg dose level will be followed to determine the progression free survival at 4 months.

#### **PHASE II**

The dose of Zotiraciclib (TG02) selected in phase I in combination with the fixed dose temozolomide will be compared to the same temozolomide dosing schedule alone in the phase II part of the study. The treatment schedule for both parts is the same. You will continue treatment until your disease gets worse, you have intolerable side effects or you have completed 12 cycles of treatment. At the time your disease worsens, if you have

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)




received temozolomide alone, you may be crossed over to receive Zotiraciclib (TG02) plus temozolomide.

Following 12 cycles of treatment, participants may continue if there is evidence of clinical benefit.

# **PRE-MEDICATIONS:**

Due to the possibility of nausea, vomiting and diarrhea with Zotiraciclib (TG02) treatment, participants will receive treatment to prevent vomiting and diarrhea before and for 24 hours following Zotiraciclib (TG02) administration. These may be tailored to the individual participant.

#### **STUDY VISITS:**

| | Screen<br>Base-<br>line | Cyc | le 1 | Сус | ele 2 | O<br>num | equent<br>odd<br>bered<br>cles | Ev<br>num | equent<br>ven<br>bered<br>cles | Off-<br>therapy |
|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | | Wk | Wk | Wk | Wk | Wk | Wk | Wk | Wk | |
| | | 2 | 4 | 2 | 4 | 2 | 4 | 2 | 4 | |
| Office visit | X | | X | | X | | X | | X | |
| Brain MRI | X | | | | X | | | | X | X |
| Blood work | X | X | X | X | X | X | X | X | X | X |
| EKG | X | | X | | X | | | | X | |
| Questionnaires* | X | | | | X | | X | | X | |
| Pregnancy<br>Test | X | | X | | X | | X | | X | X |

<sup>\*</sup> Questionnaires:

Symptom Burden Questionnaire will be done at baseline and with MRI scans.

At cycle 1, 2 and every 4 weeks:

- You will have a physical exam in NOB clinic
- You will have a pregnancy test (if appropriate) and an EKG at cycle 1, 2 and every 8 weeks

Every other week:

You will have blood collected for routine blood tests every other week

Every 8 weeks:

You will have an MRI of the brain. With each MRI:

• You will also be asked to complete a symptom burden questionnaire to

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)




determine if you have symptoms of depression, anxiety, and general well-being or function. This will take only a few minutes to complete.

### ADDITIONAL RESEARCH BLOOD AND TISSUE SAMPLES:

Research blood will be collected in the final 12 patients enrolled in Phase I at the following times: pre-dose, 1 hour, 2 hours, 4 hours, 24 hours and 48 hours after the dose. This set of blood samples will only occur in the first cycle of the protocol. Tumor sample will be needed to confirm the diagnosis before you start the study. Should you need surgery for your cancer during the study, we may collect tissue for research purposes.

# **BIRTH CONTROL**

If you are a woman who is breast feeding or pregnant, you may not take part in the study because we don't know how this medicine would affect your baby or your unborn child. If you are a woman who can become pregnant, or are the partner of a woman who can become pregnant, you will need to practice an effective form of birth control before starting study treatment, during study treatment and for 30 days after the last dose of study medication. If you think that you or your partner is pregnant, you should tell your study doctor or nurse at once

Effective forms of birth control include:

- abstinence
- intrauterine device (IUD)
- hormonal [birth control pills, injections, or implants]
- tubal ligation
- vasectomy

Other forms of birth control require the use of more than 1 method:

- Latex condom
- Diaphragm
- Cervical Cap

# RISKS OR DISCOMFORTS OF PARTICIPATION

What side effects or risks can I expect from being in this study?

While on the study, you are at risk for these side effects. You should discuss these with your doctor. There also may be other side effects that we cannot predict. Other drugs will be given to make side effects less serious and uncomfortable.

# **ZOTIRACICLIB (TG02) RISKS IN HUMANS**

# **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving Zotiraciclib (TG02), more than 20 and up to 100 may have:

- Diarrhea
- Nausea (urge to vomit)
- Vomiting
- Upset stomach
- Constipation
- Decreased appetite
- Abdominal pain
- Moderate to severe low white blood cell count

- Low potassium and phosphorus in the blood
- Shortness of breath and cough
- Elevated blood sugar
- Dizziness
- Elevated blood pressure
- Muscle aching
- Low platelet count

| OCCASIONAL, SOME MAY BE SERIOUS | |
|---|---|
| In 100 people receiving Zotiraciclib (TG02), from 4 to 20 may have: | |
| • Pneumonia | • rash |
| <ul> <li>Elevated liver enzyme</li> </ul> | • confusion |
| <ul> <li>Severe infection</li> </ul> | • fever |
| | Kidney failure |

Please tell the study doctor or study staff right away if you have any side effects. Please tell them if you have any other problems with your health or the way you feel during the study, whether or not you think they are related to the study drug.

Zotiraciclib (TG02) citrate may affect the electrical activity of the heart that coordinates the heart's beating. Medications that affect this electrical activity of the heart, taken with Zotiraciclib (TG02) citrate should be avoided. Your study doctor will make decisions about your medications on a case by case basis and discuss this with you.

You should inform the study doctor before you start any new medications, including prescription, over-the-counter, or herbal products. If you are having stomach upset, consult with your physician for recommended medications.



#### TEMOZOLOMIDE RISKS

# **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving Temozolomide, more than 20 and up to 100 may have:

- Constipation, nausea, vomiting, diarrhea
- Dizziness
- Muscle weakness, paralysis, difficulty walking
- Trouble with memory
- Tiredness
- Difficulty sleeping
- Hair loss

### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving Temozolomide, from 4 to 20 may have:

- Headache, seizure
- Infection, especially when white blood cell count is low
- Low platelet count
- Moderate to severe low white blood cell count
- Anemia which may cause tiredness
- Bruising, bleeding

## RARE, AND SERIOUS

In 100 people receiving Temozolomide, 3 or fewer may have:

- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Cancer of bone marrow caused by chemotherapy
- Damage to the bone marrow (irreversible) which may cause infection, bleeding, may require blood transfusions
- Rash
- Severe skin rash with blisters and can involve inside of mouth and other parts of the body

#### **Other Risks**

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

Questionnaires may contain questions that are sensitive in nature. You may refuse to answer any question that makes you feel uncomfortable. The primary use of the information you provide is to assess the severity of your symptoms. Submission of this information is voluntary. If you have concerns after completing the questionnaire, you are encouraged to contact your doctor or the study doctor.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)




MRI scans cannot be done on people who have a cardiac pacemaker, neural pacemaker, surgical metal clips in the brain or on blood vessels, cochlear implants, or foreign metal objects within the eye. At the time of your MRI, you will be asked about these things. When you are in the scanning machine, a feeling of claustrophobia may come over you, and there will be a repetitive thumping noise. Cool air will surround you, and the room is lit so you will not feel like you are in a cave or underground. It is important to remain still during the MRI scan. If you are very claustrophobic in MRI scanners, you may ask your physician for a mild sedative for the procedure. If you do this, you must not drive a vehicle after the MRI. You can notify the MRI technologist of any discomfort you feel. The medicine that is used for the injection may rarely (1:2000) cause an allergic reaction such as hives, shortness of breath, or low blood pressure. The medical personnel in the MRI room are prepared to treat you for this kind of reaction. The MRI study will be stopped.

This study may involve unpredictable risks to the participants.

# Risks for gadolinium enhanced MRI scans:

#### **Procedure**

During part of the MRI you will receive gadolinium, a contrast agent, through an intravenous (iv) catheter. It will be done for medical purposes.

Risks

The risks of an IV catheter include bleeding, infection, or inflammation of the skin and vein with pain and swelling.

Mild symptoms from gadolinium infusion occur in fewer than 1% of those who receive it and usually go away quickly. Mild symptoms that may occur include: coldness in the arm at injection, a metallic taste, headache, and nausea. In an extremely small number of patients, fewer than one in 300,000 people, more severe symptoms have been reported including: shortness of breath, wheezing, lowering of blood pressure. You should not receive gadolinium if you previously had an allergic reaction to it. You will be asked about such allergic reactions before gadolinium is given.

People with kidney disease are at risk for a serious reaction to gadolinium contrast called "nephrogenic systemic fibrosis (NSF)". This condition always involves the skin and can also involve the muscles, joints and internal organs. NSF has resulted in a very small number of deaths. A blood test of your kidney function may be done within the month before an MRI scan with gadolinium contrast. You will not receive gadolinium for a research MRI scan if your kidney function is below the safe level.

Most of the gadolinium contrast leaves the body in the urine. However, the FDA has issued a safety alert that indicates small amounts of gadolinium may remain in the body for months to years. The effects of the retained gadolinium are not clear. At this time, retained gadolinium has not been linked to health risks in people whose kidneys work well. Some types of gadolinium contrast drugs are less likely to remain in the body than others. In this study, we will use the gadolinium contrast drugs that are less likely to remain in the body.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)




We use gadobutrol which is a form of gadolinium contrast that is less likely to accumulate in the body than older types of gadolinium. You will receive additional information called a medication guide about the contrast medication you will receive.

Please tell your research team if you have had any MRI scans in the past 12 months. We will also give you additional information called a "Medication Guide." Upon request, we will give you individual information about retained gadolinium we see on your studies.

### POTENTIAL BENEFITS OF PARTICIPATION

# Are there benefits to taking part in this study?

The aim of this study is to determine a safe dose and to see if this experimental treatment will cause your tumors to shrink. We do not know if you will receive personal medical benefit from taking part in this study. These potential benefits could include shrinking of your tumor or lessening of your symptoms, such as pain, that are caused by the cancer. Because there is not much information about the drug's effect on your cancer, we do not know if you will benefit from taking part in this study, although the knowledge gained from this study may help others in the future who have cancer.

#### ALTERNATIVE APPROACHES OR TREATMENTS

## What other choices do I have if I do not take part in this study?

Instead of being in this study, you have these options:

- You could have a different treatment for your relapsed brain tumor. Possible alternative treatments include Optune, procarbazine, Gliadel® wafer, lomustine, carmustine, carboplatin, irinotecan, bevacizumab, etoposide. Enrolling in this trial means you will be foregoing available treatments that are approved based on studies demonstrating some clinical benefit in patients with your disease. You do not have to join this study.
- Taking part in another study
- Getting comfort care, also called palliative care. This type of care helps reduce
  pain, tiredness, appetite problems and other problems caused by the cancer. It
  does not treat the cancer directly. Instead, it tries to improve how you feel.
  Comfort care tries to keep you as active and comfortable as possible.

Please talk to your doctor about these and other options.

### STOPPING THERAPY

Your doctor may decide to stop your therapy for the following reasons:

- if he/she believes that it is in your best interest
- if your disease comes back during treatment and you cannot or choose not to cross over to TMZ+ Zotiraciclib (TG02)
- if you have side effects from the treatment that your doctor thinks are too severe

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)




- if new information shows that another treatment would be better for you
- if you become pregnant

In this case, you will be informed of the reason therapy is being stopped.

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. However, according to FDA guidelines, information collected on you up to that point may still be provided to Adastra Pharmaceuticals or designated representatives. If you withdraw your consent and leave the trial, any samples of yours that have been obtained for the study and stored at the NCI can be destroyed upon request. However, any samples and data generated from the samples that have already been distributed to other researchers or placed in the research databases cannot be recalled and destroyed.

### **Conflict of Interest**

The National Institutes of Health (NIH) reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a Protocol Review Guide. You may ask your research team for a copy of the Protocol Review Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines, but they do not need to report their personal finances to the NIH.

Members of the research team working on this study may have up to \$15,000 of stock in the companies that make products used in this study. This is allowed under federal rules and is not a conflict of interest.

Adastra Pharmaceuticals is providing the Zotiraciclib (TG02) for this study to NIH without charge. No NIH investigator involved in this study receives payments or other benefits from any company whose drug, product or device is being tested. However, there are some non-NIH collaborators on this study who may receive payments or benefits, limited by the rules of their workplace.

### COMPENSATION, REIMBURSEMENT, AND PAYMENT

# Will you receive compensation for participation in the study?

Some NIH Clinical Center studies offer compensation for participation in research. The amount of compensation, if any, is guided by NIH policies and guidelines.

You will not receive compensation for participation in this study.

# Will you receive reimbursement or direct payment by NIH as part of your participation?

Some NIH Clinical Center studies offer reimbursement or payment for travel, lodging or meals while participating in the research. The amount, if any, is guided by NIH policies and guidelines.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)




On this study, the NCI will cover the cost for some of your expenses. Some of these costs may be paid directly by the NIH and some may be reimbursed after you have paid. Someone will work with you to provide more information.

# Will taking part in this research study cost you anything?

NIH does not bill health insurance companies or participants for any research or related clinical care that you receive at the NIH Clinical Center.

- If some tests and procedures are performed outside the NIH Clinical Center, you may have to pay for these costs if they are not covered by your insurance company.
- Medicines that are not part of the study treatment will not be provided or paid for by the NIH Clinical Center.
- Once you have completed taking part in the study, medical care will no longer be provided by the NIH Clinical Center.

### CLINICAL TRIAL REGISTRATION AND RESULTS REPORTING

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

### USE OF SPECIMENS AND DATA FOR FUTURE RESEARCH

As part of this study, we are obtaining specimens and data from you. We plan to use these specimens and data for studies going on right now, as well as studies in the future. These studies may provide additional information that will be helpful in understanding brain tumors or other diseases or conditions. This could include studies to develop other research tests, treatments, drugs, or devices, that may lead to development of a commercial product by the NIH and/or its research or commercial\_partners. There are no plans to provide financial compensation to you if this happens. Also, it is unlikely that we will learn anything from these studies that may directly benefit you. By agreeing to let us use your specimens and data, you give the NIH any rights you may have in the specimens and data.

We may share your specimens and data with other researchers. They may be doing research in areas similar to this research or in other unrelated areas. These researchers may be at NIH, other research centers and institutions, or industry sponsors of research.

We will not contact you to ask about each of these future uses. These specimens and data will be stripped of identifiers such as name, address or account number, so that they may be used for future research on any topic and shared broadly for research purposes. It is also possible that the stored specimens and data may never be used. Results of research done on your specimens and data will not be available to you or your doctor. It might help people who have cancer and other diseases in the future.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)




If you do not want your stored specimens and data used for future research, please contact us in writing and let us know that you do not want us to use your specimens and/or data. Then any specimens that have not already been used or shared will be destroyed and your data will not be used for future research. However, it may not be possible to withdraw or delete materials or data once they have been shared with other researchers.

# **Genomic Data Sharing**

As part of this research study, we will put your genomic data in a large database for broad sharing with the research community. These databases are commonly called data repositories. The information in this database will include but is not limited to genetic information, race and ethnicity, and sex. If your individual data are placed in one of these repositories, they will be labeled with a code and not with your name or other information that could be used to easily identify you, and only qualified researchers will be able to access them. These researchers must receive prior approval from individuals or committees with authority to determine whether these researchers can access the data.

Summary information about all of the participants included in this study (including you) is being placed in a database and will be available through open access. That means that researchers and non-researchers will be able to access summary information about all the participants included in the study, or summary information combined from multiple studies, without applying for permission. The risk of anyone identifying you with this information is very low.

NIH policies require that genomic data be placed in a repository for sharing. Therefore, we cannot offer you a choice of whether your data will be shared. If you do not wish to have your data placed in a repository, you should not enroll in this study.

## CONFIDENTIALITY PROTECTIONS PROVIDED IN THIS STUDY

If we share your specimens or data with other researchers, in most circumstances we will remove your identifiers before sharing your specimens and data. You should be aware that there is a slight possibility that someone could figure out the information is about you.

# Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The NIH and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Institutes of Health Intramural Institutional Review Board
- Qualified representatives from Adastra Pharmaceuticals, the pharmaceutical company who produces Zotiraciclib (TG02)

When results of an NIH research study are reported in medical journals or at scientific meetings, the people who take part are not named and identified. In most cases, the NIH will not release any information about your research involvement without your written permission. However, if

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)




you sign a release of information form, for example, for an insurance company, the NIH will give the insurance company information from your medical record. This information might affect (either favorably or unfavorably) the willingness of the insurance company to sell you insurance.

Further, the information collected for this study is protected by NIH under a Certificate of Confidentiality and the Privacy Act.

# **Certificate of Confidentiality**

To help us protect your privacy, the NIH Intramural Program has received a Certificate of Confidentiality (Certificate). With this certificate, researchers may not release or use data or information about you except in certain circumstances.

NIH researchers must not share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if requested by a court.

The Certificate does not protect your information when it:

- 1. is disclosed to people connected with the research, for example, information may be used for auditing or program evaluation internally by the NIH; or
- 2. is required to be disclosed by Federal, State, or local laws, for example, when information must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA);
- 3. is for other research;
- 4. is disclosed with your consent.

The Certificate does not prevent you from voluntarily releasing information about yourself or your involvement in this research.

The Certificate will not be used to prevent disclosure to state or local authorities of harm to self or others including, for example, child abuse and neglect, and by signing below you consent to those disclosures. Other permissions for release may be made by signing NIH forms, such as the Notice and Acknowledgement of Information Practices consent.

# **Privacy Act**

The Federal Privacy Act generally protects the confidentiality of your NIH medical records we collect under the authority of the Public Health Service Act. In some cases, the Privacy Act protections differ from the Certificate of Confidentiality. For example, sometimes the Privacy Act allows release of information from your medical record without your permission, for example, if it is requested by Congress. Information may also be released for certain research purposes with due consideration and protection, to those engaged by the agency for research purposes, to certain federal and state agencies, for HIV partner notification, for infectious disease or abuse or neglect reporting, to tumor registries, for quality assessment and medical audits, or when the NIH is involved in a lawsuit. However, NIH will only release information from your medical record if it is permitted by both the Certificate of Confidentiality and the Privacy Act.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)




#### POLICY REGARDING RESEARCH-RELATED INJURIES

The NIH Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the NIH, the NIH Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.

# PROBLEMS OR QUESTIONS

If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Jing Wu, MD., <u>jing.wu3@nih.gov</u>, at 240-760-6036. You may also call the NIH Clinical Center Patient Representative at 301-496-2626, or the NIH Office of IRB Operations at 301-402-3713, if you have a research-related complaint or concern.

#### CONSENT DOCUMENT

Please keep a copy of this document in case you want to read it again.




| | have read the explanation about this study and questions. I consent to participate in this study. | have been given the |
|---|---|---|
| Signature of Research Participant | Print Name of Research Participant | Date |
| about this study and have been<br>authorized to make research deci<br>authority to provide consent to thi | ive (LAR) for an Adult Unable to Consent: I have given the opportunity to discuss it and to ask quesions on behalf of the adult participant unable to a study. As applicable, the information in the above consent who agrees to participate in the study. | estions. I am legally consent and have the |
| Signature of LAR | Print Name of LAR | Date |
| Investigator: | | |
| Signature of Investigator | Print Name of Investigator | Date |
| | <b>Onsent process only:</b> This section is only required if y lish consent form has been approved by the IRB for u | _ |
| Signature of Witness* | Print Name of Witness | Date |
| An interpreter, or other incompactificated | CTION TO BE COMPLETED REGARDING dividual, who speaks English and the participant's and served as a witness. The investigator obtain | s preferred language |
| PATIENT<br>IDENTIFICATION | <b>Consent to Participate in a Clinical Research Stu</b><br>NIH-2977 (4-17) | dy |

Version Date: 06/01/2020


File in Section 4: Protocol Consent (2) IRB NUMBER: 17C0009 IRB APPROVAL DATE: 07/07/2020

| ١ | <b>AFD</b> I | CAL | RECC | RD |
|------|--------------|-----|------|------|
| - 17 | , , , , , , | | | ,,,, |

CONSENT TO PARTICIPATE IN AN NIH CLINICAL RESEARCH STUDY

| An interpreter, or other indi | vidual, who speaks | English and the | participant's prefer | red language |
|---|---|---|---|---|
| facilitated | | | | |
| the administration of informed cons | ent but <u>did not</u> serve | as a witness. The n | ame or ID code of th | e person |
| providing interpretive support is: | | | | |


